CLINICAL TRIAL: NCT06749535
Title: The Detection of Chronic Obstructive Pulmonary Disease in Patients With Diabetes Mellitus
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHS/Batch-Spring23/039
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: group 1 — The aim of my study, we should diagnose diabetes on time. If diabetes mellitus untreated or uncontrolled for a long they directly affect all over the body, mostly they caused chronic disease due to hyperglycemia that damages the blood vessels. Rapture or damages the blood vessels of the lung causes COPD.

SUMMARY:
"Background: Chronic obstructive pulmonary disease (COPD) is an ongoing lung condition caused by damage to the lungs. The damage results in swelling and irritation, also called inflammation, inside the airways that limit airflow into and out of the lungs. Diabetes can worsen the progression and prognosis of COPD.

DETAILED DESCRIPTION:
If inflammation cause in lungs breathing process become disturbed. If damages the air sacs (alveoli) that cause emphysema. COPD mainly starts with asymptomatic patients who do not realize that they have it. It mostly affects older people or middle-aged. Its symptoms become develop slowly but with the time they become worsen, patient change their life style and treatment become helpful to prevent from chronic disease The Detection of Chronic Obstructive Pulmonary Disease in Patients with Diabetes Mellitus.

Methods: The Study design was cross sectional and carried out in hospital, Lahore from July 2024 to Jan 2024. All eligible patients who were Diabetes Mellitus in the study through random sampling technique.

ELIGIBILITY:
Inclusion Criteria:

* Age: 30-65 years Gender: Both
* Male and female
* At least 5-10 year history of Diabetes Mellitus
* Chronic Obstructive Pulmonary Disease

Exclusion Criteria:

* Patients who smoke prolong.
* Patient having other diseased (asthma, lung carcinoma).
* Patients having Acute Respiratory Distress Syndrome (ARDS)."

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Aim is to access the Chronic Obstructive Pulmonary Disease in Patients With Diabetes Mellitus
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-03-02 (Estimated)

PRIMARY OUTCOMES:
copd | 12 Months
  The aim of my study, we should diagnose diabetes on time. If diabetes mellitus untreated or uncontrolled for a long they directly affect all over the body, mostly they caused chronic disease due to hyperglycemia that damages the blood vessels. Rapture or damages the blood vessels of the lung causes COPD.

CONTACTS AND LOCATIONS:
Locations (1):
- Gulab devi hospital, Ferozepur Rd, Nishtar Town, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No